CLINICAL TRIAL: NCT03904602
Title: EdemaWear to Reduce Edema in Hospitalized Patients With Chronic Venous Insufficiency: A Pilot Study
Brief Title: EdemaWear to Reduce Edema in Hospitalized Patients With CVI:
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients experienced translocation of edema from lower extremities to trunk heightening concern about triggering congestive heart failure in frail elders.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Virginia Capasso, Clinical Nurse Specialist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018 JIE
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Chronic Venous Insufficiency
Keywords: Chronic Venous Insufficiency; CVI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Edema Wear (Experimental): Edema Wear fuzzy wale compression garment worn on lower extremities continuously for 5 days or until discharge if less than 5 days.
  Interventions: Device: Edema Wear fuzzy wale compression garment

INTERVENTIONS:
Device: Edema Wear fuzzy wale compression garment — net-like compression structure of Lycra spandex elastic yarn with longitudinal fuzzy wales (similar to corduroy fabric)

SUMMARY:
The purpose of this pilot study is to evaluate the effectiveness of EdemaWear® fuzzy wale longitudinal compression stockings on reducing lower extremity edema in hospitalized adult patients with a history of CVI who are at high risk of consequent venous leg ulcers (VLU) and patient experience with continuously wearing Edema Wear for up to five days

DETAILED DESCRIPTION:
Hospitalized patients with chronic venous insufficiency (CVI) are at high risk of venous leg ulcers (VLU) due to lower leg edema and skin changes. Since VLU are associated with prolonged morbidity and appreciable financial burden to the patient and society, prevention of VLU by reduction of lower leg edema is paramount. Although the mainstay of VLU prevention is compression, there is a gap in the acute care toolbox to manage the symptom of CVI edema. Currently, ACE bandages are the single most common 'compression wraps' stocked on inpatient units. The disadvantages of ace wraps, which are long-stretch bandages, are two-fold: 1) lower working pressure impeding venous return to the heart, and 2) higher resting pressure that may cause a tourniquet effect and consequent tissue ischemia. A newer moderately-priced mild compression product (15-20 mmHg), EdemaWear® longitudinal elastic compression stockinet, offers an alternative for hospitalized patients. There is limited evidence about the effectiveness of EdemaWear® (that is, modest reduction of lower leg edema) derived from one case series and two comparative evaluations involving only patients in out-patient clinics. This pilot study will expand the evidence related to the effectiveness of EdemaWear® in reducing lower leg edema to include hospitalized patients with CVI. .

The proposed pilot interventional study which involves a single-group repeated measures design with mixed methods has three aims:

1. evaluate the effectiveness of EdemaWear fuzzy wale elastic compression stockinet in reducing lower extremity edema in hospitalized adult patients with chronic venous insufficiency as measured by the difference in the volume of each lower extremity from Day 1 and Day 5 of data collection or the day of discharge if it occurs in less than five days
2. determine through interviews the experience of patients continuously wearing EdemaWear compression garment for up to five days or hospital discharge if it occurs in less than five days
3. qualitatively describe nurses' perceptions of their patients experience with continuously wearing EdemaWear compression garment for up to five days or hospital discharge if it occurs in less than five days

The procedure:

* Initial data collection related to demographic variables (age, gender, race, ethnic background), primary diagnosis, comorbid conditions (Charlson Comorbidity Index), CEAP classification of chronic venous disease, medication / treatment regimen, degree of lower extremity edema, volume of lower leg peripheral pulses, ankle-brachial indexes
* Daily data collection related to changes in health status and treatment
* Daily measurement of the girth of both lower extremities at 10 cm intervals from mid-foot, up the legs, to just below the knees.
* Daily interviews of patient and nursing staff related to experience of continuously wearing EdemaWear for up to five days or hospital discharge if it occurs in less than five days

Data analysis:

- Descriptive statistics will be performed on demographic and physiological variables, including number / percent for nominal variables and mean (+SD) for continuous variables. Data will be analyzed to decide whether they meet the assumptions of the planned analyses. Repeated measures ANOVA will be used to determine whether there are significant differences in the volume of the lower legs treated with EdemaWear® across the five time periods. The alpha level will be set at p < .05.

Qualitative data from daily interviews of patients and nursing staff will be analyzed by

* the PI and Co-Is of this study. Content analysis will be used to analyze the data. The unit of analysis will be phrases or sentences contained in responses to questions in the Interview Guides. Content Analysis is a qualitative research method that is used to isolate and interpret themes, issues, and repeated patterns. They refine understanding as new insights about the data emerge. The strategies for analysis outlined by Downe - Wamboldt will be followed.

ELIGIBILITY:
Inclusion Criteria:

* history of CVI (Clinical classification 1-5), with > 2+ edema of the lower legs,
* > 2+ peripheral pulses (popliteal, dorsalis pedis [DP], and posterior tibial [PT]) or audible biphasic / triphasic Doppler signal, if pulses not palpable.

Exclusion Criteria:

* open venous stasis ulcer(s) or other wounds on lower legs
* lymphedema or risk factors for lymphedema
* acute heart failure with active management
* known deep vein thrombosis (DVT) with subtherapeutic anticoagulation
* peripheral arterial disease (PAD) with reduced / absent pulses
* known or suspected inferior vena caval (IVC) compression
* circumference of lower leg < 45 cm or > 115 cm (size limits of small and extra-large EdemaWear®)
* severely altered mental status or lacking capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
change in lower leg volume | up to 5 days
  Difference between volume of lower leg / foot between Day 1 and Day 5 (or day of hospital discharge if less than 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Capasso, PhD, APRN, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lal BK. Venous ulcers of the lower extremity: Definition, epidemiology, and economic and social burdens. Semin Vasc Surg. 2015 Mar;28(1):3-5. doi: 10.1053/j.semvascsurg.2015.05.002. Epub 2015 May 8. PMID 26358303
- [Background] O'Donnell TF Jr, Passman MA, Marston WA, Ennis WJ, Dalsing M, Kistner RL, Lurie F, Henke PK, Gloviczki ML, Eklof BG, Stoughton J, Raju S, Shortell CK, Raffetto JD, Partsch H, Pounds LC, Cummings ME, Gillespie DL, McLafferty RB, Murad MH, Wakefield TW, Gloviczki P; Society for Vascular Surgery; American Venous Forum. Management of venous leg ulcers: clinical practice guidelines of the Society for Vascular Surgery (R) and the American Venous Forum. J Vasc Surg. 2014 Aug;60(2 Suppl):3S-59S. doi: 10.1016/j.jvs.2014.04.049. Epub 2014 Jun 25. No abstract available. PMID 24974070
- [Background] Eberhardt RT, Raffetto JD. Chronic venous insufficiency. Circulation. 2014 Jul 22;130(4):333-46. doi: 10.1161/CIRCULATIONAHA.113.006898. No abstract available. PMID 25047584
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Brodovicz KG, McNaughton K, Uemura N, Meininger G, Girman CJ, Yale SH. Reliability and feasibility of methods to quantitatively assess peripheral edema. Clin Med Res. 2009 Jun;7(1-2):21-31. doi: 10.3121/cmr.2009.819. Epub 2009 Feb 26. PMID 19251582
- [Background] Gogalniceanu P, Lancaster RT, Patel VI. Clinical Assessment of Peripheral Arterial Disease of the Lower Limbs. N Engl J Med. 2018 May 3;378(18):e24. doi: 10.1056/NEJMvcm1406358. No abstract available. PMID 29719182
- [Background] Bailey MA, Griffin KJ, Scott DJ. Clinical assessment of patients with peripheral arterial disease. Semin Intervent Radiol. 2014 Dec;31(4):292-9. doi: 10.1055/s-0034-1393964. PMID 25435653
- [Background] Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, Fowkes FG, Hiatt WR, Jonsson B, Lacroix P, Marin B, McDermott MM, Norgren L, Pande RL, Preux PM, Stoffers HE, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Epidemiology and Prevention; Council on Clinical Cardiology; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012 Dec 11;126(24):2890-909. doi: 10.1161/CIR.0b013e318276fbcb. Epub 2012 Nov 16. No abstract available. PMID 23159553
- [Background] Sibley RC 3rd, Reis SP, MacFarlane JJ, Reddick MA, Kalva SP, Sutphin PD. Noninvasive Physiologic Vascular Studies: A Guide to Diagnosing Peripheral Arterial Disease. Radiographics. 2017 Jan-Feb;37(1):346-357. doi: 10.1148/rg.2017160044. Epub 2016 Sep 30. PMID 27689831
- [Background] Casley-Smith JR. Measuring and representing peripheral oedema and its alterations. Lymphology. 1994 Jun;27(2):56-70. PMID 8078362
- [Background] Latchford S, Casley-Smith JR. Estimating limb volumes and alterations in peripheral edema from circumferences measured at different intervals. Lymphology. 1997 Dec;30(4):161-4. No abstract available. PMID 9476247
- [Background] Downe-Wamboldt B. Content analysis: method, applications, and issues. Health Care Women Int. 1992 Jul-Sep;13(3):313-21. doi: 10.1080/07399339209516006. PMID 1399871
- See also: Bjork R. The long and short of it: Understanding compression bandaging. Wound Care Advisor. 2013; 2(6). — https://woundcareadvisor.com/best-practices-vol2-no6/
- See also: EdemaWear® New Compression Textile. — https://compressiondynamics.com/
- See also: numeric-pain-rating-scale — https://www.sralab.org/rehabilitation-measures/